CLINICAL TRIAL: NCT04422561
Title: Use of Ivermectin as a Prophylactic Option in Asymptomatic Family Close Contact for Patient With COVID-19
Brief Title: Prophylactic Ivermectin in COVID-19 Contacts
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Waheed Shouman, professor of chest diseases, Zagazig University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: ZU-IRB#6150/31-5-2020
Record Dates: First submitted 2020-06-06; First posted 2020-06-09 (Actual); Results first posted 2020-08-27 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: COVID
MeSH Terms: interventions — Ivermectin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ivermectin group (Experimental): Contacts who will receive prophylactic ivermectin
  Interventions: Drug: Ivermectin Tablets
- Control group (No Intervention): Contacts who will be only observed without prophylaxis

INTERVENTIONS:
Drug: Ivermectin Tablets — two doses 72 hours apart
  Arms: Ivermectin group

SUMMARY:
asymptomatic family close contact of confirmed COVID -19 patient will receive prophylactic ivermectin and will be followed up for 14 days for any symptoms & diagnosis of COVID -19

ELIGIBILITY:
Inclusion Criteria:

family contact of confirmed COVID-19 case

Exclusion Criteria:

* refuse to participate and receive the drug pregnancy or lactation known hypersensitivity to ivermectin

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2020-05-31 (Actual); Primary Completion 2020-07-14 (Actual); Study Completion 2020-07-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig University, Zagazig, Sharqia Province, Egypt

RESULTS

PARTICIPANT FLOW:
Groups:
- Ivermectin Group: Contacts who will receive prophylactic ivermectin
  Ivermectin Tablets:
  40-60 kg (15mg/day) 60-80kg (18mg/day) >80kg (24mg/day)
Period: Overall Study
Arm/Group | Ivermectin Group | Control Group
Started | 228 | 112
Completed | 203 | 101
Not Completed | 25 | 11
Not completed — Lost to Follow-up | 25 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ivermectin Group | Control Group | Total
Number analyzed (Participants) | 203 | 101 | 304
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.75 (14.93) | 37.69 (16.95) | 38.72 (15.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 51 | 148
  Male | 106 | 50 | 156
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Development of Symptoms ( Fever ,Cough, Sore Throat, Myalgia,Diarrhea, Shortness of Breath)
Description: history taking and clinical examination
Time Frame: within 14 days after enrollement
Measure: Count of Participants; unit: Participants
Arm/Group | Ivermectin Group | Control Group
Number analyzed (Participants) | 203 | 101
Participants | 15 | 59

2. Secondary Outcome: Development of COVID
Description: by swab
Time Frame: within 14 days after enrollement
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 14 days
Arm/Group | Ivermectin Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/203 | 0/101
Serious Adverse Events (participants affected / at risk) | 0/203 | 0/101
Other Adverse Events (participants affected / at risk) | 11/203 | 0/101
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ivermectin Group (N=203) | Control Group (N=101)
nausea (Gastrointestinal disorders) | 2 | 0
diarrhea (Gastrointestinal disorders) | 3 | 0
burning sensation (Gastrointestinal disorders) | 1 | 0
tingling/numbness (Nervous system disorders) | 1 | 0
heart burn (Gastrointestinal disorders) | 1 | 0
abdominal pain (Gastrointestinal disorders) | 1 | 0
sleepiness (Nervous system disorders) | 1 | 0
fatigue (General disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-31): https://cdn.clinicaltrials.gov/large-docs/61/NCT04422561/Prot_SAP_000.pdf